CLINICAL TRIAL: NCT02421718
Title: Standard Follow-up Program (SFP) for Lung Cancer Patients Treated With Radiotherapy or Chemoradiation
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SFP LUNG
Record Dates: First submitted 2015-04-07; First posted 2015-04-21 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: Acute toxicity; Late toxicity; Prediction models
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiotherapy
  Other Names: Chemoradiation

SUMMARY:
Motive:

In order to improve the treatment technique, a comprehensive follow-up program is needed to obtain all relevant patient, treatment and toxicity data from lung cancer patients.

Goal:

To set-up and maintain a database containing treatment results in terms of tumor control, side effects, complications and patient-reported quality of life.

A standard database of patients receiving photon treatment will be created. These data are then linked to dose-volume data of radiotherapy, with the aim to build prediction models for both tumor control and toxicity after radio (chemo) therapy that can later be used for selecting patients for proton treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NSCLC or SCLC-LD or thymoma or lung metastases (treated with stereotactic radiotherapy)
* Patients receiving radiotherapy dose > 40 Gy

Exclusion Criteria:

* Failure to comply with any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Non-Small Cell Lung Cancer (NSCLC) or Small Cell Lung Cancer - Limited Disease (SCLC-LD) or thymoma or lungmetastases (treated with stereotactic radiotherapy), receiving radiotherapy dose > 40 Gy.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-03; Primary Completion 2025-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | Highest during and within 2 weeks after last day of radiation therapy
  esophagitis (Common Terminology Criteria for Adverse Events, version 4.0)
Late toxicity | Highest within one year after last day of radiation therapy
  esophagitis (Common Terminology Criteria for Adverse Events, version 4.0); pneumonitis (Common Terminology Criteria for Adverse Events, version 4.0)

SECONDARY OUTCOMES:
Overall survival | at 1 year after first day of radiation therapy
Overall survival | at 2 years after first day of radiation therapy
Overall survival | at 3 years after first day of radiation therapy
Overall survival | at 4 years after first day of radiation therapy
Overall survival | at 5 years after first day of radiation therapy
Loco-regional tumor control | at 1 year after first day of radiation therapy
Loco-regional tumor control | at 2 years after first day of radiation therapy
Loco-regional tumor control | at 3 years after first day of radiation therapy

OTHER OUTCOMES:
Patient-rated symptoms and Quality-of-Life | Within 1 week before or after last day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at 3 months after first day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at 6 months after first day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at one year after first day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at 2 years after first day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at 3 years after first day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at 4 years after first day of radiation therapy
Patient-rated symptoms and Quality-of-Life | at 5 years after first day of radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Robin Wijsman, MD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands